CLINICAL TRIAL: NCT02517086
Title: Vascular Changes Due to Different Treatments of Lymphedema Secondary to Postoperative Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Monique Silva Rezende, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HC-FMRP nº 810616/2014
Record Dates: First submitted 2015-06-10; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Lymphedema
Keywords: blood circulation
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- therapeutic exercises (Active Comparator): The applied therapeutic exercises involve shoulder movements including flexion, extension, abduction, adduction, internal and external rotation in isolated or combined movements, with ten repetitions of each movement, associated with the music, and stretching movements finalizing the sequence of movements.
  Interventions: Other: therapeutic exercises
- elastic compression (Active Comparator): exercises for upper limb will be performed for an hour associated with the use of elastic compression. Elastic compression will be effected through a clamp brand compression of 30-40 mmHg according to the measures of voluntary member.
  Interventions: Other: elastic compression
- functional compressive bandaging (Active Comparator): exercises for upper limb will be performed for an hour associated with the use of functional compressive bandaging. The functional compressive bandaging will be held with the volunteer sitting with ipsilateral upper limb resting on the support surgery. After hydration member a cotton mesh is used to prevent friction density 1cm strip of foam on the member to be wrapped. Elastic bandages of cotton will be involved 5 cm, 10 cm, 15 cm from the fingers to the axillary region multilayered
  Interventions: Other: functional compressive bandaging

INTERVENTIONS:
Other: therapeutic exercises — The applied therapeutic exercises involve shoulder movements including flexion, extension, abduction, adduction, internal and external rotation in isolated or combined movements, with ten repetitions of each movement, associated with the music, and stretching movements finalizing the sequence of movements.
  Arms: therapeutic exercises
Other: elastic compression — exercises for upper limb will be performed for an hour associated with the use of elastic compression. Elastic compression will be effected through a clamp brand compression of 30-40 mmHg according to the measures of voluntary member.
  Arms: elastic compression
Other: functional compressive bandaging — exercises for upper limb will be performed for an hour associated with the use of functional compressive bandaging. The functional compressive bandaging will be held with the volunteer sitting with ipsilateral upper limb resting on the support surgery. After hydration member a cotton mesh is used to prevent friction density 1cm strip of foam on the member to be wrapped. Elastic bandages of cotton will be involved 5 cm, 10 cm, 15 cm from the fingers to the axillary region multilayered
  Arms: functional compressive bandaging

SUMMARY:
The objective of this study is to evaluate the effect of elastic compression, functional compressive bandaging (ECF) and active exercises in the bloodstream of the upper member ipsilateral to the surgical procedure for the treatment of breast cancer.

DETAILED DESCRIPTION:
With increasing survival of women treated for breast cancer, it becomes necessary to evaluate the effect of therapeutic resources in morbidity due to surgical treatment of breast cancer. The objective of this study is to evaluate the effect of elastic compression, functional compressive bandaging (ECF) and active exercises in the bloodstream of the upper member ipsilateral to the surgical procedure for the treatment of breast cancer. The study will be conducted according to design random cross over and wash out period of 7 days. They will be evaluated 30 volunteers aged between 45 and 70 years, submitted to treatment of breast cancer. The volunteers will be submitted to three different therapeutic procedures applied randomly by lot: active exercises, functional compressive bandaging with active exercises and elastic compression with active exercises. The profile of blood flow, including speed and direction, will be assessed by Doppler ultrasound before and after, at 0, 15, 30 minutes. Normality will be verified by the Shapiro-Wilk test, and the effect of behavior between pre- and post-intervention will be evaluated by ANOVA two-way followed by post-hoc test Friedman followed rank, p <0.05 . The data obtained in the study are intended to enhance the forms of physical therapy intervention in the face of circulatory morbidities resulting from breast cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with breast cancer undergoing surgical treatment combined with axillary dissection or sentinel node biopsy
* diagnosed with moderate to severe unilateral lymphedema

Exclusion Criteria:

* Women with muscle-tendon injury and / or joint damage in the -affected limb,
* skin disorders,
* diabetes,
* circulatory disease not controlled, -chemotherapy
* radiotherapy,
* diagnostic with metastasis in the upper limb
* women pregnancy.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Doppler Ultrasound- velocity of blood flow | one day
  Doppler ultrasound is used to measure the velocity of blood flow of the axillary and brachial vein of the upper limb with lymphedema

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Guirro, Principal Investigator — University of Sao Paulo- Ribeirao Preto- Brazil